CLINICAL TRIAL: NCT07092865
Title: A Phase 2b, Non-randomized, Controlled, Open-label, Extension Study to Evaluate the Persistence of Immune Response of the Adjuvanted RSVPreF3 Vaccine and the Safety and Immunogenicity Following Revaccination in Lung and Kidney Transplant Recipients (>=18 Years of Age)
Brief Title: A Study Evaluating Persistence of the Immune Response of the Adjuvanted Respiratory Syncytial Virus (RSV) Vaccine and the Safety and Immune Response Following Revaccination in Adults 18 Years of Age and Above Who Received Lung or Kidney Transplant
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 224083; 2024-519730-23-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2025-07-23; First posted 2025-07-30 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus (RSV); Adjuvated RSVPreF3 vaccine; Solid organ transplant (SOT); Kidney SOT; Lung SOT; Immunocompromised (IC) patients; Humoral immune response; Safety; Reactogenicity
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IC Revaccination Group (Experimental): Lung or kidney transplant recipients undergoing chronic immunosuppressive therapy who received 1 and 2 doses of the adjuvanted RSVPreF3 vaccine (IC_1 and IC_2 groups respectively) in the RSV OA=ADJ-023 parent study will receive a revaccination dose of adjuvanted RSVPreF3 vaccine at Visit 1 (Day 1) in the current study.
  Interventions: Biological: Adjuvanted RSVPreF3 vaccine

INTERVENTIONS:
Biological: Adjuvanted RSVPreF3 vaccine — 1 dose of adjuvanted RSVPreF3 vaccine administered intramuscularly at Visit 1 (Day 1).

SUMMARY:
This study evaluates persistence of the immune response of the adjuvanted RSV vaccine and the safety and immunogenicity following revaccination in adults 18 years of age and above who received lung or kidney transplant.

DETAILED DESCRIPTION:
Lung or kidney transplant recipients undergoing chronic immunosuppressive therapy, who received 1 (IC_1 group) and 2 (IC_2 group) doses of the adjuvanted RSVPreF3 vaccine in the RSV OA=ADJ-023 study [parent study; NCT05921903], will receive an additional dose of the adjuvanted RSVPreF3 vaccine in the current study. As pre-assigned in protocol, the participants that received 1 dose and 2 doses of adjuvanted RSVPreF3 vaccine in the parent study will be analysed separately in the current study for the immune response analyses, and under an overall group (IC Revaccination group) for the demographic and safety analyses.

ELIGIBILITY:
Inclusion Criteria:

* Participants of the RSV OA=ADJ-023 study from the Per Protocol Set (Visit 3 for participants in IC_1 and Visit 4 for participants in IC_2 group), who received either 1 or 2 doses of the adjuvanted RSVPreF3 vaccine and for whom the immunogenicity data are available.
* Participants who, can and will comply with the requirements of the protocol (e.g., completion of the paper diary cards (as applicable), return for follow-up visits, ability to access and utilize a phone or other electronic communications, have regular contact to allow evaluation during the study).
* Written or witnessed informed consent obtained from the participant prior to performance of any study-specific procedure.
* Female participants of nonchildbearing potential may be enrolled in the study. Non childbearing potential is defined as hysterectomy, bilateral oophorectomy, bilateral salpingectomy, and post-menopause.
* Female participants of childbearing potential may be enrolled in the study if the participant:
* has practiced adequate contraception from 1 month prior to study intervention administration, and
* agreed to continue adequate contraception until 1 month after study intervention, and
* has a negative pregnancy test on the day of and prior to study intervention administration.
* Participant who has received an ABO compatible allogeneic kidney or lung transplant (allograft) more than 12 months (365 days) prior to the study intervention administration.
* Participant receiving maintenance immunosuppressive therapy for the prevention of allograft rejection.

Specific inclusion criteria for kidney transplant (KTx) patients

• Participant with stable kidney function, stability defined as less than 20% variability between last two results of eGFR or in the opinion of the investigator after investigator review of more than the last two results of eGFRs and based on medical history.

Specific inclusion criteria for lung transplant (LTx) patients • Participant with stable lung function, with stability defined as the stability in the FEV1 compared to post-transplant baseline FEV1 and based on medical history of the last 3 months, in the opinion of the investigator.

Exclusion Criteria:

Medical conditions

* Any history of dementia or any medical condition that moderately or severely impairs cognition.
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study (e.g., life-threatening disease likely to limit survival up to study end).
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention
* Acute or chronic clinically significant cardiovascular or hepatic functional abnormality, as determined by physical examination or laboratory screening tests.
* Recurrent or uncontrolled neurological disorders or seizures. Participants with medically controlled chronic neurological diseases can be enrolled in the study as per investigator assessment, provided that their condition will allow them to comply with the requirements of the protocol.
* Any condition which, in the judgment of the investigator, would make IM injection unsafe.
* Any other clinical condition that might pose additional risk to the participant due to participation in the clinical study.

Prior/Concomitant therapy

* Vaccination with RSV-antigen containing vaccine after 1 or 2 doses received in the RSV OA=ADJ-023 study.
* Use of any investigational or non-registered product (drug, vaccine, or medical device) other than the study intervention administration during the period beginning 30 days before the study intervention administration (Day -30 to Day 1), or their planned use during the study period (up to Month 12).
* Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the study intervention administration and ending 30 days after the study intervention administration*. In the case of COVID-19 and inactivated/subunit/split influenza vaccines, this time window can be decreased to 14 days before and after study intervention administration.

  * If emergency mass vaccination for an unforeseen public health threat (e.g., a pandemic) is recommended and/or organized by the public health authorities outside the routine immunization program, the time period of 30 days described above can be reduced, if necessary for that vaccine, provided it is used according to the local governmental recommendations and that the Sponsor is notified.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/invasive medical device).

Other exclusion criteria

* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
* Any study personnel or their immediate dependents, family, or household members.
* Planned move during the study period that will prohibit participating in the study until study end.
* Pregnant or lactating female participant.
* Female participant planning to become pregnant or planning to discontinue contraceptive precautions.
* More than one organ transplanted (i.e., kidney-liver or kidney-other organ(s) transplanted). Dual organ is allowed (double kidney or double lung).
* History of events that, in the opinion of the investigator, may put the participant at increased risk for chronic allograft dysfunction.
* Participant with an episode of allograft rejection within 3 months (90 days) prior to Visit 1.
* Histologic evidence of chronic allograft injury.
* Active treatment for acute rejection.
* Current diagnosis of malignancy (except non-melanoma skin cancer that does not require systemic therapy).
* Any autoimmune conditions or pIMDs that in the opinion of the investigator may put the participant at increased risk.
* Any confirmed or suspected HIV infection or primary immunodeficiency disease or ongoing CMV infection with a viremia > 200 IU/mL.
* Use of anti-CD20 or other B-cell monoclonal antibody agents (e.g., rituximab) as induction, maintenance and/or therapeutic immunosuppressive therapy for the prevention of allograft rejection within 9 months (274 days) prior to Visit 1.
* Use of investigational and non-registered immunosuppressants at the local/country level, unless specifically prescribed for the prevention of allograft rejection, and which are non-registered and:
* available locally through compassionate use programs,
* submitted for and pending local/country registration,
* approved and registered for use in other countries with well-documented SmPC or Prescribing Information. The name of the active component(s) of these immunosuppressants must be provided in the concomitant medication listing.
* Evidence or high suspicion, in the opinion of the investigator, of noncompliance or nonadherence to use of induction and/or maintenance immunosuppressive therapies.
* Any clinically significant (based on the Investigator's clinical judgement) hematologic (hemoglobin level, white blood cell, lymphocyte, neutrophil, eosinophil, platelet red blood cell count and erythrocyte mean corpuscular volume) and/or biochemical (ALT, AST, creatinine, blood urea nitrogen) laboratory abnormality.

Specific exclusion criteria for KTx patients:

* Previous allograft loss secondary to recurrent primary kidney disease. Multiple consecutive kidney transplants are allowed if the reason for a previous allograft loss is not recurrent primary kidney disease.
* Evidence of significant proteinuria/albuminuria in the opinion of the investigator.

Specific exclusion criteria for LTx patients:

* At study intervention administration visit, diagnosis of documented acute pulmonary infection within the 2 prior weeks, based on the following: clinical, radiological, and/or physiological deterioration; OR isolation of an organism from a clinically relevant BAL fluid culture.
* Patients with diagnosis of chronic lung allograft dysfunction, defined as a decrement of 20% or more in FEV1 compared to post-transplant baseline FEV1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2027-01-12 (Estimated); Study Completion 2027-07-16 (Estimated)

PRIMARY OUTCOMES:
RSV-A neutralizing titers expressed as Geometric mean titers (GMTs) | At Visit 1 (Day 1) of the current study
  RSV-A neutralizing titers are given as GMTs and are expressed as Estimated Dilution 60 (ED60). GMT is calculated by taking the anti-log of the mean of the log titer transformations.
RSV-B neutralizing titers expressed as GMTs | At Visit 1 (Day 1) of the current study
  RSV-B neutralizing titers are given as group GMTs and are expressed as ED60. GMT is calculated by taking the anti-log of the mean of the log titer transformations.
RSV-A neutralizing titers expressed as Mean geometric increase (MGI) | At Visit 1 (Day 1) of the current study over 30 days post last dose in the RSV OA=ADJ-023 study
  MGI is defined as the geometric mean of the within participant ratios of two timepoints (ie., ratio of titers observed at Visit 1 over titers observed 30 days post last dose in the RSV OA=ADJ-023 parent study).
RSV-B neutralizing titers expressed as MGI | At Visit 1 (Day 1) of the current study over 30 days post last dose in the RSV OA=ADJ-023 study
  MGI is defined as the geometric mean of the within participant ratios of two timepoints (ie., ratio of titers observed at Visit 1 over titers observed 30 days post last dose in the RSV OA=ADJ-023 parent study).
RSV-A neutralizing titers expressed as GMTs | At Visit 2 (Day 31) of the current study
  RSV-A neutralizing titers are given as GMTs and are expressed as ED60. GMT is calculated by taking the anti-log of the mean of the log titer transformations.
RSV-B neutralizing titers expressed as GMTs | At Visit 2 (Day 31) of the current study
  RSV-B neutralizing titers are given as GMTs and are expressed as ED60. GMT is calculated by taking the anti-log of the mean of the log titer transformations.
RSV-A neutralizing titers expressed as GMTs | At Visit 3 (Day 180) of the current study
  RSV-A neutralizing titers are given as GMTs and are expressed as ED60. GMT is calculated by taking the anti-log of the mean of the log titer transformations.
RSV-B neutralizing titers expressed as GMTs | At Visit 3 (Day 180) of the current study
  RSV-B neutralizing titers are given as GMTs and are expressed as ED60. GMT is calculated by taking the anti-log of the mean of the log titer transformations.

SECONDARY OUTCOMES:
GMT ratio of RSV-A neutralizing titers | At Visit 1 (Day 1) of the current study
  RSV-A neutralizing titers are given as group GMTs and are expressed as ED60. GMT is calculated by taking the anti-log of the mean of the log titer transformations.
GMT ratio of RSV-B neutralizing titers | At Visit 1 (Day 1) of the current study
  RSV-B neutralizing titers are given as group GMTs and are expressed as ED60. GMT is calculated by taking the anti-log of the mean of the log titer transformations.
RSV-A neutralizing titers expressed as MGI | At Visit 2 (Day 31) over Visit 1 (Day 1) and at Visit 3 (Day 180) over Visit 1 (Day 1) [each visit of the current study]
  MGI is defined as the geometric mean of the within participant ratios of two timepoints (ie., ratio of titers observed at Visit 2 over titers observed at Visit 1, and Visit 3 over Visit 1).
RSV-B neutralizing titers expressed as MGI | At Visit 2 (Day 31) over Visit 1 (Day 1) and at Visit 3 (Day 180) over Visit 1 (Day 1) [each visit of the current study]
  MGI is defined as the geometric mean of the within participant ratios of two timepoints (ie., ratio of titers observed at Visit 2 over titers observed at Visit 1, and Visit 3 over Visit 1).
RSV-A neutralizing titers expressed as MGI | At Visit 2 (Day 31) of the current study over 30 days post last dose in the RSV OA=ADJ-023 study
  MGI is defined as the geometric mean of the within participant ratios of two timepoints (ie., ratio of titers observed at Visit 2 over titers observed at 30 days post last dose in the RSV OA=ADJ-023 parent study).
RSV-B neutralizing titers expressed as MGI | At Visit 2 (Day 31) of the current study over 30 days post last dose in the RSV OA=ADJ-023 study
  MGI is defined as the geometric mean of the within participant ratios of two timepoints (ie., ratio of titers observed at Visit 2 over titers observed at 30 days post last dose in the RSV OA=ADJ-023 parent study).
Number of participants reporting each solicited administration site event | Visit 1 (Day 1 [day of revaccination]) to Day 7 of the current study
  Solicited administration site events assessed are pain, redness and swelling.
Number of participants reporting each solicited systemic event | Visit 1 (Day 1 [day of revaccination]) to Day 7 of the current study
  Solicited systemic events assessed are fever, headache, myalgia (muscle pain), arthralgia (joint pain) and fatigue (tiredness).
Number of participants reporting unsolicited adverse events (AEs) | Visit 1 (Day 1 [day of revaccination]) to Day 30 of the current study
  An unsolicited AE is an AE that was either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events. Unsolicited AEs include both serious and nonserious AEs.
Number of participants reporting any serious adverse events (SAEs) | Visit 1 (Day 1 [day of revaccination] to Visit 3 (Day 180) of the current study
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, is considered or defined as an important medical event, or abnormal pregnancy outcomes. Any SAE = occurrence of the SAE regardless of relation to study vaccination.
Number of participants reporting related SAEs and fatal SAEs | Visit 1 (Day 1 [day of revaccination] to study end (Day 365) of the current study
  Related SAE = SAE assessed by the investigator as related to the study vaccination. Fatal SAE = occurrence of a fatal SAE regardless of relation to study vaccination.
Number of participants reporting any Potential immune-mediated disease (pIMDs) and related pIMDs | Visit 1 (Day 1 [day of revaccination] to study end (Day 365) of the current study
  pIMDs are a subset of Adverse events of special interest (AESIs) that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology. Any pIMDs = occurrence of the pIMDs regardless of relation to study vaccination. Related pIMDs = pIMDs assessed by the investigator as related to the study vaccination.
Number of participants reporting AESIs specific to kidney and lung SOT patients | Visit 1 (Day 1 [day of revaccination] to study end (Day 365) of the current study
  AESIs specific to kidney and lung SOT patients include signs of transplant/allograft rejection.

CONTACTS AND LOCATIONS:
Locations (24):
- United States (6):
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Temple, Texas
- GSK Investigational Site, Herston, Queensland, Australia
- Canada (3):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Toronto, Ontario
- GSK Investigational Site, Giessen, Germany
- Italy (2):
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Pavia
- Japan (5):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Seoul, South Korea
- Spain (5):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santander

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf